CLINICAL TRIAL: NCT02193165
Title: The Comparative Efficacy of Three Oral Hygiene Multi-component Regimens Encompassing the Use of a Manual Toothbrush, Toothpaste and a Mouthwash in Controlling Established Dental Plaque and Gingivitis.
Brief Title: The Clinical Efficacy of Three Oral Hygiene Regimens Using a Manual Toothbrush, Toothpaste and a Mouthwash in Controlling Dental Plaque and Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2014-07-PG-REG-PR-BS
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen 1 (Active Comparator): triclosan/fluoride toothpaste + cetylpyridinium chloride Mouthwash
  Interventions: Drug: triclosan/fluoride toothpaste + cetylpyridinium chloride Mouthwash
- Regimen 2 (Active Comparator): stannous fluoride toothpaste + cetylpyridinium chloride Mouthwash
  Interventions: Drug: stannous fluoride toothpaste + cetylpyridinium chloride Mouthwash
- Regimen 3 - Control group (Placebo Comparator): fluoride toothpaste + fluoride Mouthwash
  Interventions: Drug: fluoride toothpaste + fluoride Mouthwash

INTERVENTIONS:
Drug: triclosan/fluoride toothpaste + cetylpyridinium chloride Mouthwash — Brush whole mouth with Total toothpaste for 1 minute, 2 times/day for 6 weeks (study duration) using a Total 360 toothbrush. Immediately after each toothbrushing, rinse whole mouth with 20 ml of mouthwash for 30 seconds.
  Other Names: Total toothpaste; Total Mouthwash
  Arms: Regimen 1
Drug: stannous fluoride toothpaste + cetylpyridinium chloride Mouthwash — Brush whole mouth with Crest Pro-Health toothpaste for 1 minute, 2 times/day for 6 weeks (study duration) using an Oral B Pro-Health toothbrush. Immediately after each toothbrushing, rinse whole mouth with 20 ml of Crest Pro-Health Multi-Protection mouthwash for 30 seconds.
  Other Names: Crest Pro-Health toothpaste; Crest Pro-Health Multi-Protection Mouthwash
  Arms: Regimen 2
Drug: fluoride toothpaste + fluoride Mouthwash — Brush whole mouth with Crest Cavity Protection toothpaste for 1 minute, 2 times/day for 6 weeks (study duration) using an Oral B Indicator toothbrush. Immediately after each toothbrushing, rinse whole mouth with 20 ml of Crest Pro-Health For Me Breezy Mint mouthwash for 30 seconds.
  Other Names: Crest Cavity Protection toothpaste; Crest Pro-Health For Me Breezy Mint mouthwash
  Arms: Regimen 3 - Control group

SUMMARY:
The objective of this clinical research study is to assess the efficacy of three oral hygiene multi-component regimens encompassing the use of a manual toothbrush, toothpaste and a mouthwash in controlling established dental plaque and gingivitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages 21-70, inclusive.
2. Availability for the six-week duration of the study.
3. Good general health.
4. Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
6. Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
7. Signed Informed Consent Form.

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removable dentures.
3. Tumor(s) of the soft or hard tissues of the oral cavity.
4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
5. Five or more carious lesions requiring immediate restorative treatment.
6. Use of antibiotics any time during the one month prior to entry into the study.
7. Participation in any other clinical study or test panel within the one month prior to entry into the study.
8. Pregnant women or women who are breast feeding.
9. Dental prophylaxis received in the past two weeks prior to baseline examinations.
10. History of allergies to oral care/personal care consumer products or their ingredients.
11. On any prescription medicines that might interfere with the study outcome.
12. An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
13. History of alcohol or drug abuse

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Comercial Plaza Trujillo, Trujillo Alto, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment at clinical site
Pre-assignment Details: There is no wash-out period prior to product randomization and distribution. Each subject was randomized and given a study treatment to follow after successfully completing the study screening procedures.
Period: 4 Week Product Use
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Started | 40 | 40 | 40
Completed | 39 (1 subject failed to keep appointments and didn't return to clinical site) | 39 (1 subject failed to keep appointments and didn't return to clinical site) | 39 (1 subject failed to keep appointments and didn't return to clinical site)
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Period: 6 Week Product Use
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Started | 39 | 39 | 39
Completed | 39 | 38 (1 subject failed to keep appointment time and didn't return to clinical site.) | 39
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 38 | 39 | 116
  >=65 years | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 14 | 47
  Male | 23 | 24 | 26 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 40 | 40 | 40 | 120
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Scores
Description: Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 3.33 (0.52) | 3.19 (0.53) | 3.31 (0.48)
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3 - Control Group; Means and standard deviations. 1 factor ANOVA to balance treatment groups to show no difference between groups. Baseline groups are balanced and baseline scores for each intervention group should not be significantly different. Significance will be determined by p<0.5; Test type: Superiority or Other; p = 0.434, ANOVA

2. Primary Outcome: Dental Plaque Scores
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Number analyzed (Participants) | 39 | 39 | 39
units on a scale | 2.78 (0.56) | 2.79 (0.52) | 3.34 (0.48)
Statistical Analysis 1: Comparison: Regimen 2 vs Regimen 3 - Control Group; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline. Significant differences between groups determined by P<0.05; Test type: Superiority or Other; p < 0.001, ANCOVA — 1 factor ANCOVA to determine difference between groups with baseline as covariate. The F statistic is used to determine significance. If significance is found then a Tukey's multiple comparison is done

3. Primary Outcome: Dental Plaque Scores
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Number analyzed (Participants) | 39 | 38 | 39
units on a scale | 2.42 (0.62) | 2.59 (0.58) | 3.38 (0.49)
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3 - Control Group; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline. Significant differences between groups will be determined at P<0.05; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Primary Outcome: Gingivitis Scores
Description: Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 1.40 (0.31) | 1.40 (0.32) | 1.44 (0.37)
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3 - Control Group; Means and standard deviations. 1 factor ANOVA to balance treatment groups to show no difference between groups. The null hypothesis states that there is no difference between groups. Differences will be noted at P<0.05. Baseline groups are balanced and baseline scores for each intervention group should not be significantly different; Test type: Superiority or Other; p = 0.816, ANOVA

5. Primary Outcome: Gingivitis Scores
Description: as for outcome 4
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Number analyzed (Participants) | 39 | 39 | 39
units on a scale | 1.19 (0.23) | 1.30 (0.27) | 1.44 (0.37)
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3 - Control Group; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline. Significant differences between intervention groups will be determined @ P<0.05; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

6. Primary Outcome: Gingivitis Scores
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Number analyzed (Participants) | 39 | 38 | 39
units on a scale | 1.03 (0.14) | 1.21 (0.24) | 1.46 (0.36)
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3 - Control Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Duration of study
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 - Control Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No